CLINICAL TRIAL: NCT01446315
Title: Assessing Decision Maker Tools for Asthma: the Asthma APGAR
Acronym: Asthma APGAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Olmsted Medical Center (Other)
Responsible Party: Principal Investigator, Barbara P. Yawn, MD, MSc, Director of Research, Olmsted Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HS018431 (AHRQ)
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Asthma
Keywords: asthma; asthma care system; effectiveness; primary care; practice based research network
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthma APGAR (Experimental): Use of new asthma care tools. Primary care practices will be provided and educated about the Asthma APGAR tool system to guide asthma care. The practices will adopt this system for all people in their practices with asthma. Outcomes will be assessed only for those who meet enrollment criteria and sign informed consent.
  Interventions: Behavioral: Use of Asthma APGAR system and tools
- Usual care (Placebo Comparator): Usual asthma care as provided by the sites.
  Interventions: Behavioral: Asthma APGAR tools

INTERVENTIONS:
Behavioral: Use of Asthma APGAR system and tools — Practices will use the Asthma APGAR control questionnaire and the care algorithm.
  Arms: Asthma APGAR
Behavioral: Asthma APGAR tools — Usual care
  Arms: Usual care

SUMMARY:
Asthma is a common problem among US adults and children. Unfortunately many people with asthma continue to suffer from asthma symptoms that could be control with better asthma care and more attention to details such as triggers, and adherence. To date the only tools available and recommended by groups such as the national asthma guideline group consider only asthma burden and do not include information on the most common factors that adversely affect asthma control. This study provides one half of the enrolled primary care offices with the Asthma APGAR which is a system of patient completed questions and a care flow sheet. The other half of the enrolled practices will continue to provide "usual" care without the support of the Asthma APGAR system. The research questions is whether or not asthma control and asthma related quality of life will be improved in people with asthma who are cared for in the intervention practices that use the Asthma APGAR system.

DETAILED DESCRIPTION:
Since this is a practice intervention study, the practices are randomized and all patients enrolled within each practice receive either the intervention based care or the usual care.

The primary outcome is asthma related quality of life obtained from patient report. Other outcomes include asthma control, also a patient reported outcome, and number of exacerbations which is obtained from patient medical record review.

ELIGIBILITY:
Inclusion Criteria:

1. Have physician diagnosed asthma
2. Male or female between ages 5 through 60 years
3. Have persistent asthma as assessed by daily use of "controller" medication
4. Receive continuity care at practice where enrolled.
5. Not have been in ICU for asthma ever
6. Do not require daily or every other day oral steroids for asthma control

Exclusion Criteria:

1. Cannot read and speak English
2. Child refuses assent

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Asthma Quality of Life Questionnaire (AQLQ) | 12 months
  Chagne in asthma relted quality of life from basline (enrollment date) to 12 months later

SECONDARY OUTCOMES:
Asthma Control Questionnaire | 12 months
  Change in asthma control from baseline to 12 month follow up.
Exacerbation rate | 12 months
  Number of emergency department visits, hospitalization and episodes of oral steroid bursts--all related to asthma, during the 12 months of follow as obtained from patient report and medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara P Yawn, MD MSc, Principal Investigator — Olmsted Medical Center
Locations (1):
- Olmsted Medical Center, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Yawn BP, Wollan PC, Rank MA, Bertram SL, Juhn Y, Pace W. Use of Asthma APGAR Tools in Primary Care Practices: A Cluster-Randomized Controlled Trial. Ann Fam Med. 2018 Mar;16(2):100-110. doi: 10.1370/afm.2179. PMID 29531100
- [Derived] Rank MA, Bertram S, Wollan P, Yawn RA, Yawn BP. Comparing the Asthma APGAR system and the Asthma Control Test in a multicenter primary care sample. Mayo Clin Proc. 2014 Jul;89(7):917-25. doi: 10.1016/j.mayocp.2014.02.016. Epub 2014 May 5. PMID 24809759